CLINICAL TRIAL: NCT00109603
Title: A Pilot Study to Determine the Impact on Dyslipidemia of the Addition of Tenofovir to Stable Background Antiretroviral Therapy in HIV-Infected Subjects
Brief Title: Effect of Tenofovir Disoproxil Fumarate on Lipid Levels in HIV Infected Adults on Stable Anti-HIV Drug Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTG A5206
Record Dates: First submitted 2005-04-29; First posted 2005-05-02 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections; Dyslipidemia; Hyperlipidemia; Hypercholesterolemia; Hypertriglyceridemia
Keywords: Treatment Experienced; TDF
MeSH Terms: conditions — HIV Infections; Dyslipidemias; Hyperlipidemias; Hypercholesterolemia; Hypertriglyceridemia | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate

SUMMARY:
The purpose of this study is to determine the effect of the anti-HIV drug tenofovir disoproxil fumarate (TDF) on lipid levels in HIV infected adults on stable anti-HIV drug therapy.

Study hypothesis: The addition of TDF to stable background antiretroviral therapy in HIV infected individuals with dyslipidemia will result in a reduction of non-HDL after 12 weeks of treatment.

DETAILED DESCRIPTION:
Use of highly active antiretroviral therapy (HAART) has resulted in significant reductions in morbidity and mortality among HIV infected people. However, significant adverse effects, including dyslipidemia, have been associated with HAART. Dyslipidemia may cause elevations in serum total cholesterol, low-density lipoprotein (LDL) cholesterol, and triglyceride concentrations, as well as a decrease in high-density lipoprotein (HDL) concentrations. Dyslipidemia is of particular concern for patients receiving HAART because the condition is associated with increased risk for cardiovascular events. TDF is an antiretroviral that has exhibited favorable lipid effects in several studies in HIV infected people, but the mechanism for the observed lipid-lowering effect of TDF is unknown. This study will evaluate the efficacy of TDF on lowering non-HDL in HIV infected adults currently on stable HAART. HAART itself will not be provided by this study.

This study will last 32 weeks. Participants will be randomly assigned to one of two study arms. Arm A participants will receive 12 weeks of TDF daily, 4 weeks of no TDF, 12 weeks of placebo daily, then 4 weeks of no TDF. Arm B participants will receive 12 weeks of placebo daily, 4 weeks of no TDF, 12 weeks of TDF daily, then 4 weeks of no TDF. Participants will continue to take their currently prescribed stable HAART regimen for the duration of the study. There will be 13 study visits over the 32 weeks of the study. Clinical assessments will occur at all visits; blood and urine collection will occur at most visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* HIV viral load less than 400 copies/ml within 28 days prior to study entry
* Treatment with stable HAART for at least 90 days prior to study entry. Patients who have taken TDF, didanosine, unboosted atazanavir, or adefovir within 90 days prior to study entry are not eligible.
* Fasting triglycerides of 150 mg/dl or greater AND less than 1000 mg/dl within 28 days prior to study entry or fasting non-HDL cholesterol 100 mg/dl or greater AND less than 250 mg/dl within 28 days prior to study
* Hepatitis B virus surface antigen negative within 6 months prior to study entry
* Have adhered to a lipid-lowering diet and exercise program for at least 28 days prior to study screening, and willing to continue both for the duration of the study
* Willing to continue any current use of hormone replacement therapy or oral contraceptives for the duration of the study. Participants must have been on a stable dose of these medications for at least 28 days prior to study entry to be eligible.
* Willing to use acceptable means of contraception

Exclusion Criteria:

* Any lipid-lowering agents within 28 days prior to study entry
* Nephrotoxins, such as foscarnet and amphotericin B, within 28 days prior to study entry
* Systemic cancer chemotherapy within 60 days prior to study entry
* Hormonal anabolic therapies or systemic steroids within 6 months prior to study entry
* Allergy or sensitivity to the study drug or its formulation
* Uncontrolled diabetes, as defined by the protocol, within 28 days prior to study entry
* Current hypothyroidism which has been treated for less than 28 days prior to study entry
* History of coronary heart disease, known atherosclerotic disease, cerebrovascular disease, peripheral vascular disease, abdominal aortic aneurysm, or arterial blockage
* Any acute illness within 28 days prior to study entry that, in the opinion of the investigator, may interfere with the study
* Current drug or alcohol abuse that, in the opinion of the investigator, may interfere with the study
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-05; Primary Completion 2007-07 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Fasting non-HDL cholesterol at baseline and Weeks 12, 16, and 28

SECONDARY OUTCOMES:
Fasting HDL, total cholesterol, and triglycerides
direct LDL by ultracentrifugation
viral load, CD4 count, and other clinical and laboratory measures

CONTACTS AND LOCATIONS:
Overall Officials: Judith Aberg, MD, Study Chair — NYU Langone Health; Marisa Tungsiripat, MD, Study Chair — The Cleveland Clinic
Locations (20):
- United States (19):
  - University of Southern California, Los Angeles, California
  - University of California, San Diego Antiviral Research Center, San Diego, California
  - University of Colorado Health Sciences Center, Denver, Denver, Colorado
  - University of Miami, Miami, Florida
  - Indiana University Hospital, Indianapolis, Indiana
  - Methodist Hospital of Indiana, Indianapolis, Indiana
  - Wishard Hospital, Indianapolis, Indiana
  - University of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University (St. Louis), St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - NYU/Bellevue, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, Galveston, Galveston, Texas
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Dube MP, Stein JH, Aberg JA, Fichtenbaum CJ, Gerber JG, Tashima KT, Henry WK, Currier JS, Sprecher D, Glesby MJ; Adult AIDS Clinical Trials Group Cardiovascular Subcommittee; HIV Medical Association of the Infectious Disease Society of America. Guidelines for the evaluation and management of dyslipidemia in human immunodeficiency virus (HIV)-infected adults receiving antiretroviral therapy: recommendations of the HIV Medical Association of the Infectious Disease Society of America and the Adult AIDS Clinical Trials Group. Clin Infect Dis. 2003 Sep 1;37(5):613-27. doi: 10.1086/378131. Epub 2003 Aug 15. No abstract available. PMID 12942391
- [Background] Grinspoon S, Carr A. Cardiovascular risk and body-fat abnormalities in HIV-infected adults. N Engl J Med. 2005 Jan 6;352(1):48-62. doi: 10.1056/NEJMra041811. No abstract available. PMID 15635112
- [Background] Martinez E, Tuset M, Milinkovic A, Miro JM, Gatell JM. Management of dyslipidaemia in HIV-infected patients receiving antiretroviral therapy. Antivir Ther. 2004 Oct;9(5):649-63. PMID 15535403
- [Background] Mehta N, Reilly M. Atherosclerotic cardiovascular disease risk in the HAART-treated HIV-1 population. HIV Clin Trials. 2005 Jan-Feb;6(1):5-24. doi: 10.1310/HT0W-NX2N-U2BM-7LUU. PMID 15765307
- [Background] Stein JH. Managing cardiovascular risk in patients with HIV infection. J Acquir Immune Defic Syndr. 2005 Feb 1;38(2):115-23. doi: 10.1097/01.qai.0000147525.26746.07. PMID 15671795
- [Result] Tungsiripat M, Kitch D, Glesby MJ, Gupta SK, Mellors JW, Moran L, Jones L, Alston-Smith B, Rooney JF, Aberg JA. A pilot study to determine the impact on dyslipidemia of adding tenofovir to stable background antiretroviral therapy: ACTG 5206. AIDS. 2010 Jul 17;24(11):1781-4. doi: 10.1097/QAD.0b013e32833ad8b4. PMID 20495438